CLINICAL TRIAL: NCT06110351
Title: Acute Clinical Outcomes of Hemorrhagic Myocardial Infarction
Acronym: MIRON-ACUTE
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine
Other Study IDs: 19978a
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute clinical outcomes 1. Mortality 2. Arrhythmia 3. Readmission 4. CVA 5. ADHF

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years of age
2. Primary PCI
3. Post-PCI cardiac biomarker labs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary PCI STEMI patients having post-PCI biomarkers
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-days and 6 months
  Prevalence of acute mortality

SECONDARY OUTCOMES:
Acute heart failure | 30-days and 6 months
  Prevalence of acute heart failure
Arrhythmia | 30-days and 6 months
  Prevalence of acute arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- IU Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No